CLINICAL TRIAL: NCT02716038
Title: A Single-arm, Phase II Study of Neoadjuvant MPDL3280A, Nab-paclitaxel and Carboplatin (MAC) in Resectable Non-small Cell Lung Cancer (NSCLC)
Brief Title: Neoadjuvant MPDL3280A, Nab-paclitaxel and Carboplatin (MAC) in NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Genentech, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ3153
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MPDL3280A, Carboplatin, Nab-paclitaxel (Experimental): Subjects with advanced or recurrent cancers receiving:
  * MPDL3280A every 21 days for up to 84 days
  * Carboplatin every 21 days for up to 84 days
  * Nab-paclitaxel every 7 days for up to 84 days
  Interventions: Drug: MPDL3280A; Drug: Carboplatin; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: MPDL3280A — MPDL3280A is a human, Fc optimized, monoclonal antibody directed against the protein ligand programmed cell death-1 ligand 1 (PD-L1), with potential immune checkpoint inhibitory and antineoplastic activities. Atezolizumab binds to PD-L1, blocking its binding to and activation of its receptor programmed death 1 (PD-1) expressed on activated T-cells, which may enhance the T-cell-mediated immune response to neoplasms and reverse T-cell inactivation. MPDL3280A 1200 mg will be administered as a 60 minute IV infusion on first administration, then over 30 minutes subsequently if tolerated.
  Other Names: Atezolizumab; RG7446
Drug: Carboplatin — Carboplatin is a second-generation platinum compound with a broad spectrum of antineoplastic properties. Carboplatin contains a platinum atom complexed with two ammonia groups and a cyclobutane-dicarboxyl residue. This agent is activated intracellularly to form reactive platinum complexes that bind to nucleophilic groups, thereby inducing intrastrand and interstrand DNA cross-links, as well as DNA-protein cross-links. These carboplatin-induced DNA and protein effects result in apoptosis and cell growth inhibition. Carboplatin area under the curve (AUC)=6 will be administered as a 30 minute IV infusion immediately after nab-paclitaxel.
  Other Names: Paraplatin; Paraplatin-Aqueous (AQ)
Drug: Nab-paclitaxel — Nab-paclitaxel is an albumin-stabilized nanoparticle formulation of the natural taxane paclitaxel with antineoplastic activity. Nab-paclitaxel binds to and stabilizes microtubules, preventing their depolymerization and so inhibiting cellular motility, mitosis, and replication. Nab-paclitaxel 100 mg/m2 will be administered as a 30 minute IV infusion.
  Other Names: Abraxane

SUMMARY:
This is a research study to test the effectiveness of nab-paclitaxel + carboplatin + MPDL3280A for treatment of non-small-cell lung carcinoma (NSCLC), which is a type of lung cancer. The study aims to determine if chemotherapy combined with immune-based therapy can lead to improvement in tumor response rates over historical response rates with chemotherapy alone.

DETAILED DESCRIPTION:
Lung cancer is the most common cancer in both men and women worldwide, accounting for 13% of incident cancers. In 2015, it was estimated there would be 221,200 new lung cancers diagnosed in the United States, with 158,040 lung cancer deaths. Approximately 85% of all lung cancers are characterized as non-small cell lung cancer (NSCLC).

Repeated studies have shown neoadjuvant cytotoxic chemotherapy to be safe prior to surgical resection of NSCLC with no difference in extent of surgical procedures performed, operative morbidity and mortality. The debate remains as to whether neoadjuvant or adjuvant chemotherapy is the best approach, with advantages and disadvantages to each.

The investigators propose that new therapies such as immune checkpoint inhibitors that demonstrate promising clinical activity in the advanced disease setting must be incorporated into the neoadjuvant setting, in order to maximize benefit early in a patient's treatment course, and with a suitable surrogate endpoint that can be used to establish a preliminary efficacy signal, prior to initiation of a large confirmatory study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed non-small cell lung cancer, of either squamous or non-squamous histology.
* Stage 1B-3A
* Deemed surgically resectable by a thoracic surgeon
* Age ≥ 18 years
* Radiologically measurable disease, as defined by response evaluation criteria in solid tumours (RECIST) v1.1
* Ability to understand and the willingness to sign a written informed consent document
* Females of child-bearing potential must:

  * Either commit to true abstinence from heterosexual contact, or agree to use, and be able to comply with, effective contraception (</=1% failure rate annually) without interruption, 28 days prior to starting therapy (including dose interruptions), and while on study medication or for a period of 90 days following treatment completion.
  * Have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy.
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following treatment discontinuation, even if he has undergone a successful vasectomy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks are preferred) or at least 10 unstained slides, with an associated pathology report, for central testing of tumor PD-L1 expression

  * Tumor tissue should be of good quality based on total and viable tumor content.
  * Patients who do not have tissue specimens meeting eligibility requirements may undergo a biopsy during the screening period.
* Adequate organ and marrow function as defined below:

  * Lymphocyte count ≥300/microliter (mcL)
  * Neutrophil count ≥1,500/mcL
  * Hemoglobin ≥9.0g/dl
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤1.5 x institutional upper limit of normal (ULN) (*Patients with Gilbert's disease: ≤3 x ULN)
  * Aspartate aminotransferase (AST)(SGOT)/alanine aminotransferase (ALT)(SGPT) ≤2.5 × ULN
  * Alkaline phosphatase ≤2.5 x ULN
  * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (*Unless the patient is on therapeutic anticoagulation)
  * Serum creatinine ≤1.5 x ULN or
  * Creatinine clearance ≥50 mL/min/1.73 m2 by Cockcroft-Gault estimation

Exclusion Criteria:

* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 5 years prior to initiation of study treatment; however, the following are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1)
* Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen (PSA) ≤ 10 mg/mL, etc.)
* Patients who are receiving any other investigational agents concurrently.
* Patients with no smoking history
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MPDL3280A, carboplatin, or paclitaxel.
* Patients with active hepatitis B or C infections or a history of HIV infection.

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen (HBsAg) test and a positive for the antibody test to detect antibodies to hepatitis B core antigen (anti-HBc) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection including tuberculosis (TB), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation (PUVA), methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1 Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Patients must not have >/= Grade 2 pre-existing peripheral neuropathy (per CTCAE)
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study
* Pregnant women
* History of interstitial lung disease or pneumonitis of any cause

Immunotherapy-Related Exclusion Criteria:

* Prior treatment with anti-PD-1, anti-CTLA-4 (cytotoxic T lymphocyte-associated antigen (CTLA-4)), or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents) within 2 weeks prior to Cycle 1, Day 1

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Shu, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pataer A, Kalhor N, Correa AM, Raso MG, Erasmus JJ, Kim ES, Behrens C, Lee JJ, Roth JA, Stewart DJ, Vaporciyan AA, Wistuba II, Swisher SG; University of Texas M. D. Anderson Lung Cancer Collaborative Research Group. Histopathologic response criteria predict survival of patients with resected lung cancer after neoadjuvant chemotherapy. J Thorac Oncol. 2012 May;7(5):825-32. doi: 10.1097/JTO.0b013e318247504a. PMID 22481232
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Langer CJ, Besse B, Gualberto A, Brambilla E, Soria JC. The evolving role of histology in the management of advanced non-small-cell lung cancer. J Clin Oncol. 2010 Dec 20;28(36):5311-20. doi: 10.1200/JCO.2010.28.8126. Epub 2010 Nov 15. PMID 21079145
- [Background] Goldstraw P, Crowley J, Chansky K, Giroux DJ, Groome PA, Rami-Porta R, Postmus PE, Rusch V, Sobin L; International Association for the Study of Lung Cancer International Staging Committee; Participating Institutions. The IASLC Lung Cancer Staging Project: proposals for the revision of the TNM stage groupings in the forthcoming (seventh) edition of the TNM Classification of malignant tumours. J Thorac Oncol. 2007 Aug;2(8):706-14. doi: 10.1097/JTO.0b013e31812f3c1a. PMID 17762336
- [Background] Pignon JP, Tribodet H, Scagliotti GV, Douillard JY, Shepherd FA, Stephens RJ, Dunant A, Torri V, Rosell R, Seymour L, Spiro SG, Rolland E, Fossati R, Aubert D, Ding K, Waller D, Le Chevalier T; LACE Collaborative Group. Lung adjuvant cisplatin evaluation: a pooled analysis by the LACE Collaborative Group. J Clin Oncol. 2008 Jul 20;26(21):3552-9. doi: 10.1200/JCO.2007.13.9030. Epub 2008 May 27. PMID 18506026
- [Background] NSCLC Meta-analyses Collaborative Group; Arriagada R, Auperin A, Burdett S, Higgins JP, Johnson DH, Le Chevalier T, Le Pechoux C, Parmar MK, Pignon JP, Souhami RL, Stephens RJ, Stewart LA, Tierney JF, Tribodet H, van Meerbeeck J. Adjuvant chemotherapy, with or without postoperative radiotherapy, in operable non-small-cell lung cancer: two meta-analyses of individual patient data. Lancet. 2010 Apr 10;375(9722):1267-77. doi: 10.1016/S0140-6736(10)60059-1. Epub 2010 Mar 24. PMID 20338627
- [Background] NSCLC Meta-analysis Collaborative Group. Preoperative chemotherapy for non-small-cell lung cancer: a systematic review and meta-analysis of individual participant data. Lancet. 2014 May 3;383(9928):1561-71. doi: 10.1016/S0140-6736(13)62159-5. Epub 2014 Feb 25. PMID 24576776
- [Derived] Shi Y, Li J, Chen M, Liu H, Ma D, Lin Y, Wang M, Xu Y. Sarcoidosis-like reaction after neoadjuvant pembrolizumab combined with chemotherapy mimicking disease progression of NSCLC induced encouraging discovery of pathological complete response. Thorac Cancer. 2021 Dec;12(24):3433-3436. doi: 10.1111/1759-7714.14228. Epub 2021 Nov 11. PMID 34761878
- [Derived] Shu CA, Gainor JF, Awad MM, Chiuzan C, Grigg CM, Pabani A, Garofano RF, Stoopler MB, Cheng SK, White A, Lanuti M, D'Ovidio F, Bacchetta M, Sonett JR, Saqi A, Rizvi NA. Neoadjuvant atezolizumab and chemotherapy in patients with resectable non-small-cell lung cancer: an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Jun;21(6):786-795. doi: 10.1016/S1470-2045(20)30140-6. Epub 2020 May 7. PMID 32386568
- See also: Howlader N, Noone AM, Krapcho M. SEER Cancer Statistics Review, 1975-2011. Based on November 2013 SEER data submission, posted to the SEER web site, April 2014. — http://seer.cancer.gov/archive/csr/1975_2011/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 patients did not continue after enrollment onto protocol regimen (7 screen fails and 1 subject withdrawal)
Period: Overall Study
Arm/Group | MPDL3280A, Carboplatin, Nab-paclitaxel
Started | 31
Completed | 26
Not Completed | 5
Not completed — Not evaluable | 1
Not completed — Not brought to surgery due to brain metastasis | 1
Not completed — Unresectable | 3

BASELINE CHARACTERISTICS:
Arm/Group | MPDL3280A, Carboplatin, Nab-paclitaxel
Number analyzed (Participants) | 31
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 2
  50-59 years | 3
  60-69 years | 12
  70-79 years | 13
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Major Pathologic Response (MPR)
Description: Major pathologic response rate (MPR) is defined as > or = 90% decrease in viable tumor.
Time Frame: 84 days
Population: 26 out of 31 enrolled participants had surgery (resectable) and evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | MPDL3280A, Carboplatin, Nab-paclitaxel
Number analyzed (Participants) | 26
Participants | 17

ADVERSE EVENTS:
Time Frame: Up to 48 months for the 31 out of the 39 enrolled/consented had continued onto protocol regimen, and 30 out of 31 had evaluable data (i.e., 1 patient determined not evaluable).
Arm/Group | MPDL3280A, Carboplatin, Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MPDL3280A, Carboplatin, Nab-paclitaxel (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 — Grade 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 — Grade 4
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MPDL3280A, Carboplatin, Nab-paclitaxel (N=30)
Neutropenia (Blood and lymphatic system disorders) | 15
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT02716038/Prot_SAP_000.pdf